CLINICAL TRIAL: NCT03001375
Title: Is it Necessary to do Splenic Flexure Mobilization in Laparoscopic Resection of Upper Rectal Tumors?
Brief Title: Laparoscopic Splenic Flexure Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abdel-samii, Lecturer of general surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6379
Record Dates: First submitted 2016-12-09; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Splenic Flexure Mobilization
Keywords: Laparoscopic colectomy.; Splenic flexure mobilization.; Anastomotic leakage.
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilization group (Active Comparator): Laparoscopic splenic flexure mobilization will be done.
  Interventions: Procedure: Laparoscopic high anterior resection splenic flexure mobilization
- Non mobilization group (Active Comparator): No mobilization of splenic flexure.
  Interventions: Procedure: Laparoscopic high anterior resection without splenic flexure mobilization

INTERVENTIONS:
Procedure: Laparoscopic high anterior resection splenic flexure mobilization
  Arms: Mobilization group
Procedure: Laparoscopic high anterior resection without splenic flexure mobilization
  Arms: Non mobilization group

SUMMARY:
This retrospective cohort study conducted on 140 patients who underwent laparoscopic anterior resection for upper rectal cancer in the period from May 2011 to November 2015, comparison will be done on splenic flexure mobilization excluding .

DETAILED DESCRIPTION:
Presently, it is acknowledged that laparoscopic colectomy for left sided colorectal cancer is the most common surgery operated in laparoscopic colorectal surgeries, However the most debatable question in such type of operations that is it mandatory to do splenic flexure mobilization or not? In the literatures colorectal surgeons divided into 2 teams, those with splenic flexure mobilization in laparoscopic left colorectal resection to have tension free, well vascularized anastomosis On the other hand those against splenic flexure mobilization reported that omitting this step does not significantly affect the leakage rate, morbidity or the oncological outcomes In this study, we evaluate the necessity of splenic flexure mobilization in laparoscopic anterior resection for upper rectal tumors and its impact on the operative time, total morbidity, leakage rate, oncological safety and continence level

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper rectal tumors.

Exclusion Criteria:

* Low and mid rectal cancer
* Splenic flexure tumors, descending colon cancer,
* patients with associated lesions in the right or transverse colon
* Emergency cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the incidence of leakage rate in laparoscopic anterior resection with splenic flexure mobilization versus non mobilization of splenic flexure | One year

IPD SHARING:
Plan to Share IPD: Undecided